CLINICAL TRIAL: NCT01927952
Title: A Prospective Randomized Comparison of Three Methods for Fixation of Hammertoes
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study withdrawn from IRB approval process by PI
Sponsor: Susan Hassenbein (Other)
Responsible Party: Sponsor-Investigator, Susan Hassenbein, Clinical Research Associate, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB - 43245
Record Dates: First submitted 2013-08-19; First posted 2013-08-23 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Acquired Deformities of Toe
Keywords: hammertoe
MeSH Terms: conditions — Hammer Toe Syndrome | interventions — Bone Wires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Kirschner wire (Active Comparator): surgical fixation using a Kirschner wire
  Interventions: Procedure: Kirschner wire
- Integra IPP-On PIP Fusion System (Active Comparator): surgical fixation utilizing the Integra IPP-On PIP Fusion System
  Interventions: Procedure: Integra IPP-On PIP Fusion System
- Stryker Smart-Toe implant (Active Comparator): surgical fixation utilizing the Stryker Smart-Toe implant
  Interventions: Procedure: Stryker Smart-Toe Implant

INTERVENTIONS:
Procedure: Kirschner wire — Surgical fixation utiliziing Kirschner wire
  Arms: Kirschner wire
Procedure: Integra IPP-On PIP Fusion System — surgical fixation utilizing the Integra IPP-On PIP Fusion System
  Arms: Integra IPP-On PIP Fusion System
Procedure: Stryker Smart-Toe Implant — surgical fixation utilizing the Stryker Smart-Toe Implant
  Arms: Stryker Smart-Toe implant

SUMMARY:
The purpose of this research project is to compare three different methods for fixation of hammertoe deformities: (1) Kirschner wire; (2) Integra IPP-ON PIP Fusion System; and (3) Stryker Smart-Toe implant.

DETAILED DESCRIPTION:
This is a prospective, randomized study and will assist us in ascertaining which of the three tested interventions has the most beneficial outcome.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (greater than or equal to 18 years of age) diagnosed with hammertoe deformity, acquired (ICD9 734.5) requiring surgical fixation
* Subject has given voluntary, written informed consent to participate in this clinical investigation.
* Subject, in the opinion of the clinical investigator, is able to understand the clinical investigation and is willing to perform all study procedures and follow-up visits
* Subject must be comfortable with speaking, reading, and understanding questions and providing responses in an available translated language.

Exclusion Criteria:

* Subjects less than 18 years of age
* Subjects with peripheral or central neurologic disease causing neurologic symptoms, including pain, dysthesia, or numbness of the operative leg
* Subjects diagnosed with complicated diabetes mellitus with noted neuropathy, diagnosed by the 10-g monofilament test
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Complications | change from baseline to 12 weeks
  Will look at number of participants with complications/adverse events including: floating toe, recurrence of hammertoe, soft tissue infection, medial/lateral mal-alignment at PIP joint, plantar flexion/hyperextension mal-alignment at DIP joint, rotation of toe and need for revision surgery.

SECONDARY OUTCOMES:
Functional Outcome | change from baseline to 12 weeks
  Will look at functional outcomes of patients as reported in the Foot and Ankle Ability Measure (FAAM) questionnaire administered to patients to assess their function pre- and post-surgery.
Patient Satisfaction | change from baseline to 12 weeks
  Will look at overall patient satisfaction with surgical care via a questionnaire administered to patients.

CONTACTS AND LOCATIONS:
Overall Officials: Umur Aydogan, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Coughlin MJ, Dorris J, Polk E. Operative repair of the fixed hammertoe deformity. Foot Ankle Int. 2000 Feb;21(2):94-104. doi: 10.1177/107110070002100202. PMID 10694020
- [Background] Reece AT, Stone MH, Young AB. Toe fusion using Kirschner wire. A study of the postoperative infection rate and related problems. J R Coll Surg Edinb. 1987 Jun;32(3):158-9. No abstract available. PMID 3656240
- [Background] Zingas C, Katcherian DA, Wu KK. Kirschner wire breakage after surgery of the lesser toes. Foot Ankle Int. 1995 Aug;16(8):504-9. doi: 10.1177/107110079501600809. PMID 8520664
- [Background] Klammer G, Baumann G, Moor BK, Farshad M, Espinosa N. Early complications and recurrence rates after Kirschner wire transfixion in lesser toe surgery: a prospective randomized study. Foot Ankle Int. 2012 Feb;33(2):105-12. doi: 10.3113/FAI.2012.0105. PMID 22381341
- [Background] Lehman DE, Smith RW. Treatment of symptomatic hammertoe with a proximal interphalangeal joint arthrodesis. Foot Ankle Int. 1995 Sep;16(9):535-41. doi: 10.1177/107110079501600904. PMID 8563920
- [Background] Caterini R, Farsetti P, Tarantino U, Potenza V, Ippolito E. Arthrodesis of the toe joints with an intramedullary cannulated screw for correction of hammertoe deformity. Foot Ankle Int. 2004 Apr;25(4):256-61. doi: 10.1177/107110070402500411. PMID 15132935
- [Background] Sarrafian SK. Correction of fixed hammertoe deformity with resection of the head of the proximal phalanx and extensor tendon tenodesis. Foot Ankle Int. 1995 Jul;16(7):449-51. doi: 10.1177/107110079501600714. PMID 7550962
- [Background] Konkel KF, Sover ER, Menger AG, Halberg JM. Hammer toe correction using an absorbable pin. Foot Ankle Int. 2011 Oct;32(10):973-8. doi: 10.3113/FAI.2011.0973. PMID 22224327
- [Background] Gadkari K, et al. A Prospective Comparison of a Permanent Intramedullary Device to K-Wire Fixation for Proximal Interphalangeal Joint Fusion: Early Results. Presented at AAOS Annual Meeting 2013, AOFAS Specialty Day
- [Background] Martin RL, Irrgang JJ, Burdett RG, Conti SF, Van Swearingen JM. Evidence of validity for the Foot and Ankle Ability Measure (FAAM). Foot Ankle Int. 2005 Nov;26(11):968-83. doi: 10.1177/107110070502601113. PMID 16309613